CLINICAL TRIAL: NCT00826917
Title: Use of 3D/4D Ultrasound in the Evaluation of Fetal Anomalies - The Use of Volumetry by Three Dimensional Ultrasound in the First Trimester
Brief Title: Use of 3D/4D Ultrasound in the Evaluation of Fetal Anomalies
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW07-293
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Homozygous αº-thalassemia; Hb Bart's Disease
Keywords: 3D, 2D, ultrasound, volumetry, multiplanar, VOCALTM, XI VOCALTM, fetal, gestational sac, placenta

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Objective 1: XI VOCALTM in 3D fetal volumetry measurement: group 1: multiplanar; group 2: VOCALTM; group 3: XI VOCALTM
- Objective 2: XI VOCALTM in 3D placental volumetry measurement: group 1: multiplanar; group 2: VOCALTM; group 3: XI VOCALTM
- Objective 3: Comparison between 2 ultrasound machine: 1. intramachine reliability for (i)fetal, (ii)gestational sac and (iii)placenta volumetry measurement for (a)multiplanar and (b)VOCALTM:- group 1:Accuvix; group 2:Voluson 730
  2. intermachine reliability for fetal, gestational sac and placenta volumetry measurement for (a)multiplanar and (b)VOCALTM for Accuvix and Voluson 730
- Objective 4:3D volumetry in fetuses at risk of Hb Bart's: Measurement of fetal, gestational sac and placenta volume per CRL quotient using multiplanar technique:- group 1: affected; group 2: unaffected

SUMMARY:
Volumetry measurements can be a potential clinical use as non-invasive tools in prenatal diagnosis and screening and helps to reduce the risk and complications of invasive procedures. 3DUS volumetry gives more precise results than 2DUS volumetry measurements, particularly, of irregularly shaped objects.

DETAILED DESCRIPTION:
Conventionally volume measurements can be made by using multiplanar or VOCALTM (Virtual Organ Computer-aided AnaLysis). Recently, a new technique, XI VOCALTM (eXtended Imaging VOCAL) has been described. Combined with the inversion mode, measurements for the liquid-filled structures can also be made. The potential use in clinical diagnosis and prediction of pathologies of volume measurements particularly in the first trimester are yet to be investigated.

3D ultrasound is found to be superior to 2D parameter in volumetry measurement. However, currently, there are still very few studies done to evaluate the potential use of volumetry measurement in clinical practice, especially of the validity and reproducibility of XI VOCALTM; and the variation of results obtained within different ultrasound machines. Due to the potential use of volumetry measurements in clinical practice, the accuracy in volumetry measurement is very important and the development of new technique need to be fully explored so that its benefits can be fully used for the contribution of clinical practice.

So far no research has been done to evaluate the difference in the results obtained between different ultrasound machines, in particularly for volumetry measurements. This is important because if there is no significant difference in results between difference machines, we can accumulate the results from these machines for a study, which can include a more variety of samples. Furthermore, it will be much easier to compare results of one machine with another for similar studies.

Both Voluson 730 and Accuvix have been used widely in research studies on 3D volumetry but comparison of the results obtained from these two machines have not been done. We do not know whether the results generated from one machine can be extrapolated to the other machine for clinical or research purpose. Thus more research needs to be done in this area.

Thus, this study is carried out to evaluate the potential use of the new modality of XI VOCALTM in the volumetry measurement of regular and irregular shaped objects, comparison of results obtained between different widely used machines, and the potential used of volumetry measurements in the prediction of common and important clinical pathologies such as αº-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

For objective 1 and 2 - Samples are recruited from our prenatal diagnostic clinic at Ysan Yuk Hospital between 11-14 weeks' gestation. They are those who come for routine scan and those who are referred from the general antenatal clinics of the same hospital which pregnancies are at risk of homologous alphaº thalassaemia.

For objective 3 - Recruitment are the same as above except samples are obtained from normal pregnancy.

For objective 4 - Recruitment are the same as above. However, study is divided into intervention group and control group. For the intervention group, data is collected from pregnancies at risk of of homozygous αº-thalassemia while for the control group, data is collected from normal pregnancies.

Exclusion Criteria:

* If women refuse to participate in the study
* Patients with other co-existing illnesses

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Use of XI VOCALTM in 3D fetal volumetry measurements,comparison with multiplanar and VOCALTM
     -restropective(2005-2007),30 singleton pregnancies,11-14 weeks' gestation, at risk of homozygous αº-thalassaemia.
  2. Use of XI VOCALTM in 3D placental volumetry measurements,comparison with multiplanar and VOCALTM
     -retrospective(2005-2007), 32 singleton pregnancies,11-14 weeks' gestation at risk of homologous alphaº thalassaemia.
  3. Comparison of 3DUS volumetry measurement between two models of ultrasound machine -prospective(December 2007-June 2008),30 singleton normal pregnancies,11-14 weeks' gestation.
  4. Use of 3DUS in fetal, gestational sac and placenta quotient measurement, fetuses at risk of homozygous αº-thalassemia(Hb Bart's disease) -retrospective(datasets July 2007-Dec 2008),singleton pregnancies,11-14 weeks' gestation,26 affected cases,34 unaffected cases,43 normal control.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Objective 1:The use of XI VOCALTM in 3D volumetry measurements of fetal head and trunk of fetuses from 11 to 14 weeks gestation and known volume phantoms and its comparison with the conventional multiplanar and VOCALTM technique | 18 months
  The objectives of this study are to compare (1) the reproducibility of multiplanar and the VOCALTM technique for 3DUS measurement of fetal volume with the new modality XI VOCALTM, and (2) validity of these three techniques using an in-vitro setting.
  The hypothesis of the study are (1) the results obtained from the new modality of XI VOCALTM is interchangeable with multiplanar and VOCALTM with similar number of steps used and (2) validity between XI VOCALTM is comparable to multiplanar and VOCALTM with similar number of steps used.
  We hypothesized XI VOCALTM can be used interchangeably with multiplanar and VOCALTM technique if similar number of steps are used in the measurement of regular objects such as fetal head and trunk.
Objective 2:The use of new modality of XI VOCALTM in 3D volumetry measurements of placenta from 11 to 14 weeks gestation and known volume phantoms and its comparison with the conventional multiplanar and VOCALTM technique | 18 months
  The objectives of this study are to compare (1) the reproducibility of multiplanar and the VOCALTM technique for 3DUS measurement of placenta volume with the new modality XI VOCALTM, and (2) validity of these three techniques using an in-vitro setting.
  The hypothesis of the study are (1) the results obtained from the new modality of XI VOCALTM is interchangeable with multiplanar and VOCALTM with similar number of steps used and (2) validity between XI VOCALTM is comparable to multiplanar and VOCALTM with similar number of steps used.
  We hypothesized that XI VOCALTM can be used interchangeably with the other two techniques for the volumetry measurement of irregular objects such as placenta if similar number of steps is used.
Objective 3:The use of 3DUS in the volumetry of first trimester pregnancy and in vitro study: comparison between two models of ultrasound machine | 18 months
  The objective of the present study are to compare (1) the reproducibility of these two machines for fetal, gestational sac and placenta 3D volumetry using multiplanar (1-mm interval) and Virtual Organ Computer-Aided Analysis (VOCAL)TM (30º) technique and (2) validity of these two machines using an in-vitro setting.
  Hypothesis of the study: 3D volumetry measurement of fetal, gestational sac and placenta volume of fetuses at 11 to 14 weeks' gestation with Voluson 730 is interchangeable with the measurement using Accuvix ultrasound machine.
  We hypothesized that the Accuvix machine could be used interchangeably with Voluson 730 for both multiplanar and VOCALTM for fetal, gestational sac and placenta volumetry measurement.
Objective 4:The use of 3DUS in the measurement of fetal, gestational sac and placenta quotient of fetuses at risk of homozygous αº-thalassemia (Hb Bart's disease) at 11 to 14 weeks' gestation | 18 months
  This study was carried out to evaluate the use of fetal, gestational sac and placenta volume measured by three-dimensional (3D) ultrasound in predicting fetal homozygous αº-thalassemia (Hb-Bart's disease).
  Hypothesis of the study: Measurement of 3D volume of the fetal, gestational sac and placenta quotient can be used as a useful tool as 2D parameter for the prediction of fetuses of homozygous alpha0-thalassaemia (Hb Bart's disease) at 11 to 14 weeks' gestation.
  We hypothesized that 3D volumetry measurement of the fetal, gestational sac and placenta quotient can serve as a useful tool as 2D parameter for the prediction of homozygous alpha0-thalassaemia (Hb Bart's disease) fetuses at 11 to 14 weeks' gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Bik Cheong, BSc(Hons), MMedSc, MBBS, Principal Investigator — The University of Hong Kong; Kwok Yin Leung, MBBS, FHKAM, Study Director — The University of Hong Kong
Locations (1):
- Tsan Yuk Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Leung KY, Cheong KB, Lee CP, Chan V, Tang MHY, Lau ETK. Prenatal diagnosis of homozygous α°-thalassemia: from an invasive to a noninvasive approach. Expert Reviews. 2009.4(3): 321-329.
- [Background] Leung KY, Cheong KB, Tang MHY, Chan V. Prenatal Diagnosis of Thalassaemia. JPOG. 2008. 34(1): 37-42.
- [Background] Leung KY, Cheong KB, Lee CP, Chan V, Lam YH, Tang M. Ultrasonographic prediction of homozygous alpha0-thalassemia using placental thickness, fetal cardiothoracic ratio and middle cerebral artery Doppler: alone or in combination? Ultrasound Obstet Gynecol. 2010 Feb;35(2):149-54. doi: 10.1002/uog.7443. PMID 20047196
- [Result] Cheong KB, Leung KY, Li TK, Chan HY, Lee YP, Tang MH. Comparison of inter- and intraobserver agreement and reliability between three different types of placental volume measurement technique (XI VOCAL, VOCAL and multiplanar) and validity in the in-vitro setting. Ultrasound Obstet Gynecol. 2010 Aug;36(2):210-7. doi: 10.1002/uog.7609. PMID 20201116
- [Result] Cheong KB, Leung KY, Chan HY, Lee YP, Yang F, Tang MH. Comparison of inter- and intraobserver agreement between three types of fetal volume measurement technique (XI VOCAL, VOCAL and multiplanar). Ultrasound Obstet Gynecol. 2009 Mar;33(3):287-94. doi: 10.1002/uog.6255. PMID 19248036
- [Result] Cheong KB, Leung KY, Chan HY, Chen M, Tang MHY. Comparison of volumetry fetus, gestational sac, and placenta obtained from two three- dimensional ultrasound machines. 18th World Congress on Ultrasound in Obstetrics and Gynecology. Ultrasound Obstet Gynecol. 2008; 32: 400.
- [Result] Cheong KB, Leung KY, Chan HY, Chen M, Tang MHY. Comparison of volumetry of fetus, gestational sac, and placenta in normal pregnancies obtained by two kinds of three dimensional ultrasound machines. 4th Asia Pacific Congress inMaternal Fetal Medicine. 17Th - 19th October, 2009. Macau Tower Convention and Entertainment Center, Macau, SAR China.
- [Result] Cheong KB, Leung KY, Li TK, Chan HY, Lee YP, Tang HY. Comparison of inter- and intraobserver agreement between three different types of placental volume measurement techniques (XI VOCALTM, VOCALTM and multiplanar). 13rd -17th Sept 2009. Ultrasound Obstet Gynecol. 2009. 34 (Suppl 1): 209.
- [Result] Cheong KB, Leung KY, Chan HY, Lee YP, Tang MHY. Comparison of inter- and intraobserver agreement between three different types of fetal volume measurement techniques (XI VOCALTM, VOCALTM and multiplanar). 13th Postgraduate Symposium, Li Ka Shing Faculty of Medicine, University of Hong Kong, Hong Kong, SAR China. 2008.
- [Result] KB Cheong, KY Leung, HY Chan, YP Lee, F Yang, MHY Tang. Comparison of inter- and intra-observer agreement between three different types of fetal volume measurement techniques (XI VOCAL, VOCAL, and multiplanar). 18th World Congress on Ultrasound in Obstetrics and Gynecology. Ultrasound Obstet Gynecol. 2008; 32(3):399.
- [Result] Cheong Kah-bik, Ng EHY.The use of volumetry by three-dimensional ultrasound in the first trimester. 2009. Postgraduate Thesis. The HKU Scholars Hub (thesis online).
- See also: KB Cheong, KY Leung, HY Chan, YP Lee, F Yang, MHY Tang. Comparison of inter- and intraobserver agreement between three types of fetal volume measurement technique (XI VOCALTM, VOCALTM and multiplanar). Ultrasound Obstet Gynecol 2009; 33: 287-294 — http://onlinelibrary.wiley.com/doi/10.1002/uog.6255/pdf
- See also: Leung KY, Cheong KB, Lee CP, Chan V, Lam YH, Tang M. Ultrasonographic prediction of homozygous alphaº-thalassemia using placental thickness, fetal cardiothoracic ratio and middle cerebral artery Doppler: alone or in combination? UOG — http://www.ncbi.nlm.nih.gov/pubmed/20047196
- See also: Cheong Kah-bik, Ng EHY.The use of volumetry by three-dimensional ultrasound in the first trimester. 2009. Postgraduate thesis. The HKU Scholars Hub (thesis online). — http://dx.doi.org/10.5353/th_b4357233